CLINICAL TRIAL: NCT06741306
Title: Comprehensive Assessment in a Longitudinal Study on Young Men Who Have Sex With Men Attracting to chemseX-2
Status: Recruiting | Type: Observational
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Collaborators: The US NIH through the International Epidemiology Databases to Evaluate AIDS (IeDEA) IeDEA Asia-Pacific (Unknown); amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Other Study IDs: IHRI025
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: ChemSex Users for YMSM
Keywords: ChemSex Users

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Group1 — Current chemsex users Men who have sex with men, Aged 16-35 years (defined as last chemsex used within 3 months), Able to communicate in Thai fluently.

SUMMARY:
CLYMAX is a two-phase observational study that assess multiple aspects of chemsex and young men who have sex with men (YMSM).

Phase I of the study (CLYMAX,IRB No. 0695/65) was a cross-sectional descriptive study using a mixed methods data collection (focusing on qualitative data collection) assessing multiple aspects of chemsex, including the patterns of chemsex use and the perspectives on factors influencing chemsex initiation/discontinuation, effects on physical health, mental health and social outcomes, and the necessary services for a comprehensive chemsex clinic among YMSM; and the acceptability and feasibility of developing a comprehensive chemsex clinic from the perspective of YMSM, their family members or peers, and clinic staff.

This phase II study (CLYMAX-2) will be a prospective cohort study using a quantitative data collection exploring the effectiveness of the implementation strategy of harm reduction models and consist of a larger number of YMSM, important baseline and follow-up information on multiple aspects of physical, psychological, and social harms.

ELIGIBILITY:
Inclusion Criteria:

1. Men who have sex with men
2. Aged 16-35 years
3. Current chemsex users (defined as last chemsex used within 3 months)
4. Able to read and communicate in Thai
5. Provide informed consent

Exclusion Criteria:

None

Ages: 16 Years to 35 Years | Sex: Male
Age Groups: Child, Adult
Study Population: Current chemsex users
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The study outcomes of phase II can be broadly categorized into implementation outcomes include the prevalence and incidence of physical, psychological, and social harms which will be evaluated by laboratory or self-reported assessments as follows: | 18 months
  STIs testing including HIV (either HIV self-testing or facility-based HIV testing), HCV, HBV, gonorrhea, chlamydia, and syphilis will be offered at baseline and month 6. It will be optional for participants to decide whether to undergo the testing. Behavioral risk, substance use, mental health, quality of life, and criminality assessments will be conducted at every visit. Categorical data will be summarized as frequencies and percentages, while continuous data will be summarized as means and standard deviations or medians and interquartile ranges, as appropriate. In addition to describing the cohort, mixed-effects regression models will be used to assess temporal changes in each health outcome. Linear models will be applied for continuous outcomes (such as changes in depression, anxiety, and quality of life scores), and logistic models will be used for dichotomous outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Siriporn Nonenoy, BNH,MPH, Study Chair — Institute of HIV Research and Inovation
Locations (2):
- Thailand (2):
  - Rainbow Sky Association of Thailand (RSAT), Bangkok, Bangkapi
  - Foundation for Action on Inclusion Rights (FAIR), Bangkok, Minburi

IPD SHARING:
Plan to Share IPD: Undecided